CLINICAL TRIAL: NCT03608605
Title: Role of Advanced MRI Sequences in Differentiating MS and Its Mimics
Brief Title: Advanced MRI Sequences in Multiple Sclerosis and Its Mimics
Acronym: MS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samaa Mostafa El-kossi, assisstant lecturer, Assiut University
Other Study IDs: 17200227
Record Dates: First submitted 2018-07-18; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — magnetic resonance imaging with advanced sequences including tractography,volumetry and inversion recovery

SUMMARY:
We aim to evaluate the role of conventional and advanced MRI sequences in:

1. Establishing the diagnosis of multiple sclerosis and differentiate it from its mimics.
2. Predict the prognosis and evaluate the treatment response in the first year of patients with multiple sclerosis.

DETAILED DESCRIPTION:
All patients in the study will be referred among those attend to Assuit university hospital with clinical symptoms suspicious of MS according to McDonald criteria 2017 with age range from (18-50 years old).

MRI study will be done for each patient. MRI study will be repeated for those already diagnosed as MS after starting the suitable treatment as decided by attending physician after one year to assess the efficacy of treatment and the patient prognosis.

MR imaging will be performed on a 1.5-T MR imaging unit (Siemens, Sembra medical system,German).

Prospectively completed data forms will be analyzed and compared. Statistical tests appropriate to the nature of the data will be used.

All patients will not be subjected to risk of any kind during this study. All patients' data will be confidentially kept. Approval of the ethical committee of Faculty of Medicine, Assiut University.

An informed consent will be taken from all patients included in this study.

* The research will be conducted only by scientifically qualified and trained personnel.
* The procedures included in this study have been already used in hospital and centers in and outside Egypt.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the study will be referred among those attend to Assuit university hospital with clinical symptoms suspicious of MS according to McDonald criteria 2017 with age range from (18-50 years old).

Exclusion Criteria:

* o Any general contraindication of MRI in some cases as presence of paramagnetic substance as pacemakers or in patients with claustrophobia.

  * Patient above 50 years old.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients among those attend to Assiut university hospital with clinical symptoms suspicious of MS according to McDonald criteria 2017 with age range from (18-50 years old).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
role of advanced MRI sequences in establishing the diagnosis of multiple sclerosis(MS) | baseline
  calculating the sensitivity,specificity and accuracy of diffusion tensor imaging (DTI) and dual inversion recovery(DIR) in differentiating MS from its mimics

SECONDARY OUTCOMES:
follow up of MS patients after one year of treatment | one year
  assess the degree of brain atrophy after one year mainly in the white matter and cerebral cortex using 3DT1WI